CLINICAL TRIAL: NCT04139096
Title: Genetic Susceptibility to Radiation Induced Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C 17-69
Record Dates: First submitted 2019-10-09; First posted 2019-10-25 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Neoplasms; Genetic Susceptibility; Radiation Exposure
MeSH Terms: conditions — Thyroid Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Case control on thyroid cancer occuring in a cohort of 7300 subjects treated during their childhood, mostly by radiotherapy, for a skin Angioma at Gustave Roussy, Villejuif France between 1947 and 1973.

This case control study, which is included in a larger european project, aims to investigate the DNA variant interacting with the risk of radiation induced thyroid cancer after irradiation.

The sutdy is planed to include about 30 cases and 30 controls. Matching criteria are date of birth, gender, and age at irradiation.

ELIGIBILITY:
Inclusion Criteria:

Diganosis of thyroid cancer during the followup or selected as a control matched on gender, date of birth and age at skin hemangioma diagnosis.

Exclusion Criteria:

No available adress Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of subjects treated for a skin hemangioma at Gustave Roussy Institute from 1947 to 1973, mostly by radiotherapy.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-09-22 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Number of Differentiated thyroid carcinoma | From hemangioma diagnosis to the end of the followup, in average 45 years after hemangioma diagnosis
  Number of differentiated thyroid carcinoma occuring in a cohort of subjects treated for a skin hemangioma during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Florent de Vathaire, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Gustae Roussy, Villejuif, Val de Marne, France

IPD SHARING:
Plan to Share IPD: No